CLINICAL TRIAL: NCT01371474
Title: Special Drug Use Investigation for PAXIL Tablet (Investigation in Case of Administered From 20mg/Day)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112308
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder | interventions — Paroxetine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed PAXIL: Patients with depression or in a depressed state starting PAXIL at 20 mg/day during study period
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine

SUMMARY:
The objective of this survey was to understand the safety and efficacy of PAXIL tablets ("PAXIL", hereinafter) when it was started at 20 mg/day in subjects with depression or in a depressed state.

ELIGIBILITY:
Inclusion Criteria:

* Patients with depression or in a depressed state
* Patients who start taking paroxetine at 20mg a day

Exclusion Criteria:

* Patients who have been treated with paroxetine prior to this investigation
* Patients with hypersensitivity to paroxetine
* Patients taking monoamine oxidase inhibitors (MAOIs) or within 2 weeks of stopping treatment with MAOIs
* Concomitant use in patients taking pimozide

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Japanese subjects with depression or in a depressed state who are considered appropriate to prescribe paroxetine tablet starting at 20mg/day according to the prescribing information
Sampling Method: Probability Sample
Enrollment: 1483 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 weeks
  Incidence of adverse events in Japanese subjects treated with paroxetine tablet based on prescribing information under the conditions of general clinical practice
Efficacy evaluation based on overall improvement | 12 weeks
  The investigator compared the general condition over 1 week before each clinical visit with that over 1 week before the start of treatment with PAXIL.
Efficacy evaluation based on severity by symptoms | 12 weeks
  At every clinical visit, the investigator rated each of the specified symptoms including depressed mood, loss of interests/concerns, anxiety, lack of motivation, physical symptoms, and sleep disorders.
Efficacy evaluation based on Beck Depression Inventory- Second Edition (BDI-II) | 12 weeks
  The investigator asked each subject to fill out the self-administered form of BDI-II at every clinical visit (recommended clinical visit schedule: 1, 2, 4, 8, and 12 weeks after the start of treatment).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline